CLINICAL TRIAL: NCT02158572
Title: A Single-arm, Open-label, Multicenter Phase 3 Study of the Contraceptive Efficacy, Safety and Tolerability of the AG200-15 Transdermal Contraceptive Delivery System (TCDS)
Brief Title: Efficacy, Safety and Tolerability Study of Agile AG200-15 Transdermal Contraceptive Delivery System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-CL23
Record Dates: First submitted 2014-06-04; First posted 2014-06-09 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: prevention of pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG200-15 (Experimental): AG200-15 is a transdermal delivery system designed to deliver daily hormone exposure of ethinyl estradiol (EE) and levonorgestrel (LNG)
  Interventions: Drug: AG200-15

INTERVENTIONS:
Drug: AG200-15 — Transdermal contraceptive delivery system
  Other Names: Transdermal contraceptive delivery system

SUMMARY:
Study of the efficacy of a contraceptive patch in 2100 healthy women for up to one year.

DETAILED DESCRIPTION:
AG200-15 is used in a 4-week (28-day) treatment cycle: a patch is applied and replaced every 7 days for 3 consecutive weeks, followed by a 1-week "patch-free" period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, sexually active woman at risk for pregnancy seeking to use hormonal contraception for at least 1 year
* Ability to demonstrate willingness to participate and adhere to study protocol

Exclusion Criteria:

* Known or suspected pregnancy
* Lactating women
* Anticipates use of condoms or any other form of back-up contraception during the study
* History of dermal sensitivity to medicated patches (nicotine) or to bandages, surgical tape, etc.
* Has a contraindication to combined estrogen-progestin contraceptive use
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Smoker who is 35 years old or over

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2032 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Garner, MD, MPH, Study Director — Agile Therapeutics

REFERENCES:
- [Derived] Nelson AL, Kaunitz AM, Kroll R, Simon JA, Poindexter AN, Castano PM, Ackerman RT, Flood L, Chiodo JA 3rd, Garner EI; SECURE Investigators. Efficacy, safety, and tolerability of a levonorgestrel/ethinyl estradiol transdermal delivery system: Phase 3 clinical trial results. Contraception. 2021 Mar;103(3):137-143. doi: 10.1016/j.contraception.2020.11.011. Epub 2020 Nov 28. PMID 33259782

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AG200-15
Started | 2032
Completed | 989
Not Completed | 1043

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | AG200-15
Number analyzed (Participants) | 2031
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2031
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (6.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2031
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2031

OUTCOME MEASURES:

1. Primary Outcome: Contraception Efficacy of AG200-15 in Subjects ≤ 35 Years of Age Regardless of BMI, Intent-to-treat (ITT) Dataset.
Description: The Pearl Index will serve as the primary contraceptive efficacy endpoint for evaluation of pregnancy rates for the study. Pearl Index is the number of on-therapy pregnancies times 1300 divided by the number of 28-day on-therapy cycles and is an estimate of the number of pregnancies per 100 woman-years of product use.
Time Frame: 1 year
Population: ITT population: all complete or incomplete on-therapy cycles in which intercourse occurred and no back-up contraception was used.
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | AG200-15
Number analyzed (Participants) | 1736
Pearl Index | 5.80 [4.5 to 7.2]

2. Secondary Outcome: Contraception Efficacy of AG200-15 in Subjects ≤ 35 Years of Age With BMI < 25 kg/m2, ITT Dataset
Description: Contraception efficacy of AG200-15 by Pearl Index in subjects ≤ 35 years of age with BMI < 25 kg/m2, ITT dataset. Pearl Index is the number of on-therapy pregnancies times 1300 divided by the number of 28-day on-therapy cycles and is an estimate of the number of pregnancies per 100 woman-years of product use.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | AG200-15
Number analyzed (Participants) | 684
Pearl Index | 3.5 [1.8 to 5.2]

3. Secondary Outcome: Contraception Efficacy of AG200-15 in Subjects ≤ 35 Years of Age With BMI ≥ 25 and < 30 kg/m2, ITT Dataset
Description: Contraception efficacy of AG200-15 by Pearl Index in subjects ≤ 35 years of age with BMI ≥ 25 and < 30 kg/m2, ITT dataset. Pearl Index is the number of on-therapy pregnancies times 1300 divided by the number of 28-day on-therapy cycles and is an estimate of the number of pregnancies per 100 woman-years of product use.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | AG200-15
Number analyzed (Participants) | 439
Pearl Index | 5.7 [3 to 8.4]

4. Other Pre Specified Outcome: Self-reported Skin Irritation at Application Site
Description: Self-reported skin irritation at application site was assessed using the following scoring method:
  0: None
  1. Mild
  2. Moderate
  3. Severe
Time Frame: 1 year
Population: Subjects who reported irritation at the application site.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AG200-15
Number analyzed (Participants) | 2023
Score | 1.31 (1.020)

5. Other Pre Specified Outcome: Self-reported Skin Itching at Application Site
Description: Self-reported skin itching at application site was assessed using the following scoring method:
  0: None
  1. Mild
  2. Moderate
  3. Severe
Time Frame: 1 year
Population: Subjects who reported itching at the application site
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AG200-15
Number analyzed (Participants) | 2023
Score | 1.6 (0.951)

6. Other Pre Specified Outcome: Self-reported Patch Adhesion
Description: Patch adhesion was reported using the following 5-point scoring method:
  0: ≥ 90% adhered (none to minimal lift)
  1. ≥ 75% adhered but < 90% (some edges showing lift)
  2. ≥ 50% adhered but < 75% (at least half of system lifts off)
  3. < 50% (more than half of the patch lifts off, but the patch remains attached)
  4. Patch completely detached.
Time Frame: 1 year
Population: Subjects that reported patch adhesion
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AG200-15
Number analyzed (Participants) | 2022
Score | 2.76 (1.518)

7. Other Pre Specified Outcome: Cycle Control
Description: Number of episodes of breakthrough bleeding (BTB) and/or breakthrough spotting (BTS) per cycle.
Time Frame: 1 year
Population: Subjects that reported BTB and/or BTS
Measure: Mean (Standard Deviation); unit: Episodes/cycle
Arm/Group | AG200-15
Number analyzed (Participants) | 2017
Episodes/cycle | 0.56 (0.391)

8. Secondary Outcome: Contraception Efficacy of AG200-15 in Subjects ≤ 35 Years of Age With BMI ≥ 30 kg/m2, ITT Dataset
Description: Contraception efficacy of AG200-15 by Pearl Index in subjects ≤ 35 years of age with BMI ≥ 30 kg/m2, ITT dataset. Pearl Index is the number of on-therapy pregnancies times 1300 divided by the number of 28-day on-therapy cycles and is an estimate of the number of pregnancies per 100 woman-years of product use.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | AG200-15
Number analyzed (Participants) | 612
Pearl Index | 8.6 [5.8 to 11.5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | AG200-15
All-Cause Mortality (participants affected / at risk) | 0/2031
Serious Adverse Events (participants affected / at risk) | 40/2031
Other Adverse Events (participants affected / at risk) | 627/2031
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG200-15 (N=2031)
Cholelithiasis (Hepatobiliary disorders) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Major depression (Psychiatric disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 4 (4)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Acute repiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alcohol use (Psychiatric disorders) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Multiorgan failure (General disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Oliguira (Renal and urinary disorders) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1)
Papillary thryriod cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Phenylketonuria (Congenital, familial and genetic disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 1 (1)
Heptitis (Hepatobiliary disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Small Intestine Gangrene (Infections and infestations) | 1 (1)
Substance Abuse (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG200-15 (N=2031)
Nasopharyngitis (Infections and infestations) | 116 (116)
Upper respiratory infection (Infections and infestations) | 100 (100)
Nausea (Gastrointestinal disorders) | 84 (84)
Headache (Nervous system disorders) | 72 (72)
Urinary tract infection (Infections and infestations) | 72 (72)
Sinusitis (Infections and infestations) | 54 (54)
Dysmenorrhoea (Reproductive system and breast disorders) | 47 (47)
Acne (Skin and subcutaneous tissue disorders) | 41 (41)
Weight increased (Investigations) | 41 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval by Agile Therapeutics, Inc. of any publication, including oral presentations and abstracts, utilizing data or any information from the ATI-CL23 study is required prior to publication submission.